CLINICAL TRIAL: NCT03434652
Title: Efficacy of Auricular Neurostimulation for Children and Adults With Cyclic Vomiting Syndrome: a Pilot Study
Brief Title: Auricular Neurostimulation for Cyclic Vomiting Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Katja Kovacic, Assistant Professor of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1102505-4
Record Dates: First submitted 2018-02-01; First posted 2018-02-15 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Cyclic Vomiting Syndrome; Abdominal Migraine
MeSH Terms: conditions — Familial cyclic vomiting syndrome; Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Each subject randomized to active vs sham therapy, then cross over to the other during next illness cycle
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active percutaneous neurostimulation (Active Comparator): Subject randomized to 5 days of active vs sham neurostimulation therapy during an illness cycle. With next illness cycle, each subject will cross over to the other one (active vs sham).
  Interventions: Device: Percutaneous neurostimulation
- Sham percutaneous neurostimulation (Sham Comparator): Each subject randomized to 5 days of active vs sham neurostimulation therapy during an illness cycle. With next illness cycle, each subject will cross over to the other one (active vs sham).
  Interventions: Device: Percutaneous neurostimulation

INTERVENTIONS:
Device: Percutaneous neurostimulation — Auricular percutaneous neurostimulation
  Other Names: Neuro-Stim System (NSS)-2 BRIDGE

SUMMARY:
This study evaluates the efficacy of auricular neurostimulation via an non-invasive percutaneous electrical nerve field stimulator in children and adults with cyclic vomiting syndrome.

DETAILED DESCRIPTION:
Cyclic vomiting syndrome (CVS) is an difficult to treat and debilitating functional gastrointestinal disorder. Majority of children and adults with CVS have concurrent severe abdominal pain and migraine-features, rendering them incapacitated during the vomiting cycle.

The vagus nerve carries signals of nausea, vomiting and pain between the brain and the gastrointestinal tract and is part of the autonomic nervous system. The autonomic nervous system appears to be in imbalance in patients with CVS during a vomiting cycle. By stimulating a branch of the vagus nerve in the outer ear, this study aims to improve symptoms and quality of life in both children and adults with CVS.

Subjects will be randomized to receive active vs sham (non-active) neurostimulation therapy for 5 days at the onset of a CVS cycle. They will then cross over to the other group (active vs sham) at the onset of the next CVS cycle. Subjects in a separate sub-study receive 6 weeks of active neurostimulation therapy (5 days/week). Pain, nausea, vomiting, anxiety, quality of life, potential side effects and overall symptom improvement will be monitored before and after therapy for the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Meeting Rome IV Pediatric or Adult criteria for Cyclic Vomiting Syndrome (CVS)
* Concurrent abdominal pain with CVS cycle
* English-speaking
* Lack of other explanation for symptoms
* Either predictable, 'calendar-timed' episodes or prodromal symptoms for 12-24 hours that are predictive of episodes onset

Exclusion Criteria:

* Medically complex and/or suffering from medical condition that may explain symptoms
* Taking a medication that may explain symptoms
* Significant developmental delays
* Patients treated with a new drug affecting the central nervous system within one week of enrollment
* Infection or severe dermatological condition of ear
* Stable vital signs
* No currently implanted electrical device
* For adults (and adolescents as applicable): pregnancy, severe cardiopulmonary disease, concurrent chronic marijuana use (>2 times/month over past 6 months prior to enrollment)

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Baxter Retching Faces Scale | From date of baseline assessment (therapy start date) through next 7 days for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  Daily nausea severity assessed by pictorial nausea faces scale 0-10 (0=no nausea; 10=worse possible nausea) with higher scores indicating worse outcomes (greater nausea).

SECONDARY OUTCOMES:
Numeric pain scale | From date of baseline assessment (therapy start date) through next 7 days for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  Daily pain severity assessed by numeric pain scale 0-10 (0=no pain; 10=worst possible pain) with higher scores indicating worse outcome (greater pain).
Anxiety | From date of baseline assessment (therapy start date) and day 5 of therapy for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  State-Trait Anxiety Inventory for Children and Adults
Health-Related Quality of Life | From date of baseline assessment (therapy start date) and day 5 of therapy for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  Patient Reported Outcomes Measurement Information Systems
Disability in Children | From date of baseline assessment (therapy start date) and day 5 of therapy for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  Functional Disability Inventory
Disability in Adults | From date of baseline assessment (therapy start date) and day 5 of therapy for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  Sheehan Disability Scale assessing disability and impairment on a scale 0-10 with higher scores indicating more disability. Three sub scales: 1) school/work, 2) social life and 3) family life are assessed (scale 0-10) with a total score reflecting the sum of the 3 subscales (total score range 0-30 with higher score indicating more disability).
Global symptoms | From date of baseline assessment (therapy start date) and day 5 of therapy for each cycle of therapy. Also assessed at follow-up visit 3 months after end of therapy and further follow-up visits up to 12 months after end of therapy.
  Global symptom improvement scale

CONTACTS AND LOCATIONS:
Overall Officials: Katja Kovacic, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Babygirija R, Sood M, Kannampalli P, Sengupta JN, Miranda A. Percutaneous electrical nerve field stimulation modulates central pain pathways and attenuates post-inflammatory visceral and somatic hyperalgesia in rats. Neuroscience. 2017 Jul 25;356:11-21. doi: 10.1016/j.neuroscience.2017.05.012. Epub 2017 May 17. PMID 28526575
- [Background] Miranda A, Taca A. Neuromodulation with percutaneous electrical nerve field stimulation is associated with reduction in signs and symptoms of opioid withdrawal: a multisite, retrospective assessment. Am J Drug Alcohol Abuse. 2018;44(1):56-63. doi: 10.1080/00952990.2017.1295459. Epub 2017 Mar 16. PMID 28301217
- [Background] Roberts A, Sithole A, Sedghi M, Walker CA, Quinn TM. Minimal adverse effects profile following implantation of periauricular percutaneous electrical nerve field stimulators: a retrospective cohort study. Med Devices (Auckl). 2016 Nov 3;9:389-393. doi: 10.2147/MDER.S107426. eCollection 2016. PMID 27843360
- [Derived] Karrento K, Zhang L, Conley W, Qazi Z, Venkatesan T, Simpson P, Li BUK. Percutaneous electrical nerve field stimulation improves comorbidities in children with cyclic vomiting syndrome. Front Pain Res (Lausanne). 2023 Jun 14;4:1203541. doi: 10.3389/fpain.2023.1203541. eCollection 2023. PMID 37389229